CLINICAL TRIAL: NCT01125267
Title: Promoting Adherence to Treatment in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Alex Kopelowicz, M.D., David Geffen School of Medicine at UCLA
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5R01MH064542-05 (NIH); 5R01MH064542-05 (NIH)
Record Dates: First submitted 2010-05-17; First posted 2010-05-18 (Estimated); Last update posted 2010-05-18 (Estimated); Status verified 2010-05

CONDITIONS: Schizophrenia
Keywords: medication adherence; schizophrenia; Mexican American; multifamily groups
MeSH Terms: conditions — Schizophrenia; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- multifamily group-adherence (Experimental): multifamily group treatment with a focus on improving adherence to antipsychotic medication
  Interventions: Behavioral: multifamily group-adherence
- multifamily group-standard (Active Comparator): multifamily group focused on problems identified by group participants
  Interventions: Behavioral: multifamily group-standard
- treatment as usual (No Intervention)

INTERVENTIONS:
Behavioral: multifamily group-adherence — multifamily groups held twice a month for one year focused on improving medication adherence using techniques derived from the Theory of Planned Behavior
  Arms: multifamily group-adherence
Behavioral: multifamily group-standard — multifamily groups held twice a month focused on general problem solving method
  Arms: multifamily group-standard

SUMMARY:
The project evaluates a culturally adapted, family-based intervention designed to promote treatment adherence among Mexican-Americans with schizophrenia using a randomized, controlled design in a public mental health setting. Mexican-American patients with schizophrenia and their families were randomly assigned to either: 1) one year of multi- family groups that emphasize the importance of attitudes towards adherence, subjective norms, and self-perceived and actual adherence skills in maintaining adherence, added to ongoing customary outpatient care; 2) standard multi-family groups without an emphasis on medication adherence, added to customary outpatient care; or 3) customary outpatient care only (monthly pharmacotherapy sessions and additional services as clinically needed). The study hypotheses are that subjects assigned to the adapted multi-family group would have better medication adherence, less psychiatric symptoms and fewer psychiatric hospitalizations throughout the course of the study (one year of treatment and one year of follow up) compared to the comparison conditions.

DETAILED DESCRIPTION:
As above

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of schizophrenia or schizoaffective disorder;
* Between 18 and 50 years of age;
* Of Mexican origin and speaks Spanish fluently;
* Was without antipsychotic medication without medical authorization for one continuous week in the month prior to hospitalization;
* Was living with his/her family of origin immediately preceding the inpatient stay and would return to live with his/her family after discharge; and
* The patient and at least one family member were willing to participate.

Exclusion Criteria:

* Patient on conservatorship or legal guardian status

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 174 (Actual)
Dates: Start 2003-04; Primary Completion 2007-09 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants who are Hospitalized in a Psychiatric Inpatient Unit | two years
  Psychiatric hospitalization will be monitored through the use of the Los Angeles County Department of Mental Health Management Information System. This allows for the data capture of all participants who are hospitalized in an inpatient unit anywhere in Los Angeles County throughout the two-yaer course of the study. Although the primary outcome variable is whether or not a participant has been hospitalized within a given assessment period, the number of hospitalizations and the number of days hospitalized across all assessment periods will be assessed, as well.

SECONDARY OUTCOMES:
Number of participants who are at least 80% adherent to their antipsychotic medication regimens during a particular assessment period | two years
  Multi-modal method of assessing medication adherence including pill count, pharmacy records and interviews of patient, key relative and treating psychiatrist. Using the Treatment Compliance Interview, participants will be rated as either non-adherent (less than 50% adherence), partially adherent (50%-79% adherent) or fully adherent (80% or greater).

CONTACTS AND LOCATIONS:
Overall Officials: Alex J Kopelowicz, MD, Principal Investigator — Geffen School of Medicine at UCLA
Locations (1):
- San Fernando Mental Health Center, Granada Hills, California, United States

REFERENCES:
- [Derived] Kopelowicz A, Zarate R, Wallace CJ, Liberman RP, Lopez SR, Mintz J. The ability of multifamily groups to improve treatment adherence in Mexican Americans with schizophrenia. Arch Gen Psychiatry. 2012 Mar;69(3):265-73. doi: 10.1001/archgenpsychiatry.2011.135. PMID 22393219